CLINICAL TRIAL: NCT02774577
Title: Acute Effects on Oxygen Consumption and Blood Flow After a Single Session of Whole Body Vibration
Brief Title: Oxygen Consumption After Acute Whole Body Vibration Session
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maíra F Pessoa (Other)
Responsible Party: Sponsor-Investigator, Maíra F Pessoa, Principal Investigator, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LACAP UFPernambuco
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Aged; Oxygen Consumption
Keywords: Oxygen Consumption; Aged; Whole Body Vibration
MeSH Terms: interventions — Aging

STUDY DESIGN:
Intervention Model Description: acute wbv session, measuring ergospirometric variables during protocol and blood pressure, borg exertion, borg dyspnoea, blood lactate, heart rate and SpO2 before and after protocol.
Masking Description: similar procedures for variables, collected into similar device and positioning, using a sham device, patented, witch reproduce infra-physiologic vibrations and sound like an actual vibrating platform

ARMS (1):
- healthy young and elderly (Experimental): young adults (20 to 30 years) compare to elderly (60 to 74 years)
  Interventions: Other: whole body vibration training in vibrating platform in young; Other: whole body vibration training in vibrating platform in elderly

INTERVENTIONS:
Other: whole body vibration training in vibrating platform in young
  Other Names: WBV
Other: whole body vibration training in vibrating platform in elderly
  Other Names: WBV

SUMMARY:
Noninvasive assessment of VO2 during a single session of whole body vibration and changes in blood flow caused by the acute activity.

DETAILED DESCRIPTION:
A single whole body vibration session into two groups, a young adults groups and elderly group, booth healthy, will be held with concomitant collection of VO2 consumed during the session, by MetaMax cortex. Immediately after the session, it will be checked peripheral blood flow through US surface in color Doppler mode.

ELIGIBILITY:
Inclusion Criteria:

* healthy young adults (between 20 to 30 years) and healthy elderly (between 60 to 74 years), sedentary according International Physical Activity Questionnaire.

Exclusion Criteria:

* presence of thrombosis, labyrinthitis, osteoporosis and individuals who have difficulty adapting to the assessment or training protocol.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
VO2 through the gas exchange measured by Cortex Metamax | up to 06 months
  an atoxic mask measure oxygen consumption and carbon dioxide production in ml/kg/min-1, breathe by breathe
peripheral blood Lactate | up to 06 months
  a noninvasive evaluate using an Lactimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil